CLINICAL TRIAL: NCT06254313
Title: The Role of CXCR4-expressing Neutrophils in Influenza-related Acute Respiratory Distress Syndrome
Brief Title: The Role of Cxcr4Hi neutrOPhils in InflueNza
Acronym: CHOPIN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/41
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Influenza; Acute Respiratory Distress Syndrome
Keywords: neutrophils; CXCR4; host resistance; disease tolerance
MeSH Terms: conditions — Influenza, Human; Respiratory Distress Syndrome | interventions — LRBA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Influenza-related ARDS group: Person with influenza virus infection proven by a positive polymerase chain reaction test for the influenza ARDS group. Additional tubes taken when blood is drawn during treatment, and bronchoalveolar fluid sample.
  Interventions: Other: Additional tubes and LBA
- Bacterial-related ARDS group: A person with a proven bacterial infection (105 colony-forming units/mL for tracheal aspirates and more than 104 colony-forming units/mL for BAL). Additional tubes taken when blood is drawn during treatment, and bronchoalveolar fluid sample.
  Interventions: Other: Additional tubes and LBA
- Extra-pulmonary (digestive inflammation) ARDS group: Person presenting with acute pancreatitis according to the 2013 international recommendations (typical pain, lipasemia above 3 times normal and/or abnormality on imaging).
  Or Person presenting with acute bacterial peritonitis based on a clinical diagnosis and bacteria isolated on peritoneal samples (RFE SFAR 2018). Additional tubes taken when blood is drawn during treatment, and bronchoalveolar fluid sample.
  Interventions: Other: Additional tubes and LBA

INTERVENTIONS:
Other: Additional tubes and LBA — 4 Additional tubes taken when blood is drawn during treatment : EDTA tubes and 2 citrate tubes and bronchoalveolar fluid sample (LBA)

SUMMARY:
Influenza is still responsible for more than 650,000 deaths per year worldwide and no major improvements in patients' care has been made despite 50 years of research. Especially, there is no therapeutic strategy targeting the dysregulated host response. CXCR4-expressing neutrophils seem to be involved in the rupture of host resistance. The aim of this study is thus to compare the percentage of blood CXCR4-expressing neutrophils between influenza survivors and non-survivors.

DETAILED DESCRIPTION:
Influenza is still responsible for more than 650,000 deaths per year worldwide and no major improvements in patients' care has been made despite 50 years of research. Most of severe influenza patients suffer from acute lung injury due to a dysregulated immune response. Neutrophils are involved in both host resistance and disease tolerance. Thanks to advances in technologies, the vast variety in neutrophils subpopulations has been revealed. In particular, the subpopulation of CXCR4-expressing neutrophils has been suggested to be involved in the rupture of disease tolerance in lung infections. Nevertheless, these data are from murine models and remain to be confirmed in humans. Moreover, the underlying mechanisms remain unknown as well as the place of primum movens, i.e. vascular or alveolar compartment. The aim of this study is thus to compare the percentage of blood CXCR4-expressing neutrophils between influenza survivors and non-survivors. Percentage of BAL CXCR4-expressing neutrophils will also be compared. To this aim, blood sampling and BAL within the 24 hours and at day 3 after admission to ICU, neutrophils isolation, immunostaining and flow cytometry acquisition will be performed within the 24 hours and at day 3 after admission to ICU. Mortality rate will be collected at Day 28 and Day 90.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 yo or above.
* Acute respiratory distress syndrome as defined by the Berlin classification.
* Invasive mechanical ventilation for less than 24 hours.
* Cause of ARDS:

  * Influenza infection proven by polymerase chain reaction OR
  * Bacterial infection (tracheal aspirate with more than 105 CFU/mL and BAL with more than 104 CFU/mL.
  * Pancreatitis according to the 2013 Working Group IAP/APA Acute Pancreatitis Guidelines.
  * Peritonitis according to the 2018 SFAR guidelines.
* Health insurance.
* Written informed consent from legal relative or representative.

Exclusion Criteria:

* Neutropenia (< 500/mm3)
* Neutrophils qualitative defect.
* Patient included in an interventional research assessing an immunomodulatory or antiviral drug.
* Acquired ImmunoDeficiency Syndrome.
* Contraindication to BAL:

  * Severe bronshospasm.
  * Out-of-control shock.
  * Intracranial high pressure.
  * Refractory hypoxemia (PaO2/FiO2 < 60 mmHg).
* Legal restriction: prisoners, pregnancy, legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of interest will be patients with acute respiratory distress syndrome according to the Berlin criteria.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biological | Day 1 after inclusion
  Percentage of blood CXCR4-expressing neutrophils within the 24 hours following admission to ICU for invasive mechanical ventilation.
Clinical | Day 28 after inclusion
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Edouard LHOMME, Dr, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique du CHU de Bordeaux
Locations (2):
- France (2):
  - Hopital Pellegrin, Bordeaux
  - Hopital Haut-Lévêque, Pessac